CLINICAL TRIAL: NCT02662088
Title: Laparoscopic-lavage Observational Study
Acronym: LLOS
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Alberto Arezzo, Associate Professor of Surgery, University of Turin, Italy
Other Study IDs: LLOSTUDY-1
Record Dates: First submitted 2016-01-20; First posted 2016-01-25 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Diverticulitis
MeSH Terms: conditions — Diverticulitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Laparoscopic-lavage: Patients with colonic diverticulitis submitted to laparoscopic lavage
  Interventions: Procedure: laparoscopic-lavage

INTERVENTIONS:
Procedure: laparoscopic-lavage

SUMMARY:
The purpose of this study is to collect a multi-institutional database including all relevant data regarding the surgical and clinical features of patients underwent to laparoscopic lavage for complicated colic diverticulitis. The main objectives are:

* To determine the surgical and clinical outcomes, in the short and long term.
* To compare results according to the different type of techniques, device used and manner of execution of the different surgical steps.
* To relate results of different surgeries with baseline characteristics of patients and stage of disease.

DETAILED DESCRIPTION:
The purpose of this study is to collect a multi-institutional database including all relevant data regarding the surgical and clinical features of patients underwent to laparoscopic lavage for complicated colic diverticulitis. The main objectives are:

* To determine the surgical and clinical outcomes, in the short and long term.
* To compare results according to the different type of techniques, device used and manner of execution of the different surgical steps.
* To relate results of different surgeries with baseline characteristics of patients and stage of disease.

This "ad hoc" registry will allow centers to retrospectively fill in the data of their patients; the information will be obtained from existing records, diagnostic tests and surgical intervention descriptions. Data will be collected and recorded by all institutions through a specific online shared system.

To facilitate and standardize data collection through a shared database and to ensure the safety of sensitive data, a special online computerized web system has been developed.

Investigators have to provide the required data as fully as possible; however, the lack of certain data does not preclude from sending the remaining data.

Specific aims

* Analyze general outcome
* Analyze the different techniques of laparoscopic lavage
* Analyze the different inclusion criteria
* Analyze the different follow-up

Primary outcome for this retrospective observational study is:

the success rate of laparoscopic peritoneal lavage, defined as the rate of patients alive with no need of further surgical treatment for recurrent attacks of diverticulitis.

Secondary outcomes are:

* conversion to any form of laparoscopy different from peritoneal lavage (with or without bowel resection)
* conversion to laparotomy (with or without bowel resection)
* 30 days post-operative mortality;
* 30 days post-operative surgical re-interventions rate;
* 30 days post-operative percutaneous drainage rate;
* hospital readmission rate for recurrence of diverticulitis;
* - rate of visualisation of colonic perforation during laparoscopic peritoneal lavage;
* surgical strategies used in case of detection of a colonic perforation;
* consistency, if any, of visceral adhesiolysis performed during the procedure;
* duration of follow-up
* post-lavage elective resection rate (lavage "bridge" to resection)

Eligibility Each patient is required to meet all of the inclusion criteria and none of the exclusion criteria.

Inclusion criteria Patients with colonic diverticulitis submitted to laparoscopic lavage

Exclusion criteria Patients with occasional finding of colo-rectal cancer

Data collection Patient demographics

* Year of birth
* Sex
* Body Mass Index (BMI)
* ASA score
* Haemodynamic condition (stable or unstable)
* Previous abdominal surgery
* Previous events of diverticulitis requiring ambulatory investigation or treatment
* Previous events of diverticulitis requiring hospitalization
* Abdominal CT scan before surgery (yes/no) and WSES stage (Sartelli M, Moore FA, Ansaloni L, Di Saverio S, Coccolini F, Griffiths EA, et al. A proposal for a CT driven classification of left colon acute diverticulitis. World J Emerg Surg. 2015 World 2015; 10: 3) Surgery
* Date of Operation
* Hinchey score (modified Kaiser AM, Jiang JK, Lake JP, Ault G, Artinyan A, Gonzalez-Ruiz C, Essani R, Beart RW Jr. The management of complicated diverticulitis and the role of computed tomography. Am J Gastroenterol 2005; 100: 910-917)
* Number of trocars inserted
* Quantity of lavage (cc)
* Conversion rate to any laparoscopic technique either than lavage
* Conversion rate to any type of open surgical technique
* Degree of adhesiolysis performed for searching eventual free colonic perforation (1. none, 2. lysis of weak adhesions, 3. actively searching for any collection with consistent amount of adhesiolysis)
* Identification of a free colonic perforation during the laparoscopic peritoneal lavage
* Surgical strategies used in case of detection of a colonic perforation (drainage, stitching, resection)
* Placement of intra-abdominal drain (number and location)
* Operative time
* Estimated blood loss
* Intraoperative complications
* Intraoperative death

Postoperative clinical findings

* Length of postoperative hospital stays
* Postoperative blood transfusion
* Liquid diet (POD number)
* Soft solid diet (POD number)
* Re-establishment of peristalsis (POD number)
* First pass of flatus (POD number)
* Drain removal (POD number)
* Length and type of intravenous antibiotic use
* Length of intravenous analgesic use

In-hospital postoperative complications

* Type of complication
* Re-operation for complication
* Dindo-Clavien Grade

Early and late surgery-related complications after discharge

* Date of hospitalization for diverticulitis recurrence
* Type of complication
* Death related to the complication
* Need of surgery (type of surgery)
* Need percutaneous drainage
* Need peritoneal lavage Follow-up
* Date of last follow-up visit
* post-Lap lavage elective resection rate (lavage as a "bridge" to resection)
* Indication to resection (symptoms, prophilaxys of further episodes of acute diverticulitis)

ELIGIBILITY:
Inclusion criteria Patients with colonic diverticulitis submitted to laparoscopic lavage

Exclusion criteria Patients with occasional finding of colo-rectal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Each patient is required to meet all of the inclusion criteria and none of the exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 404 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
success rate | 12 months
  the success rate of laparoscopic peritoneal lavage, defined as the rate of patients alive with no need of further surgical treatment for recurrent attacks of diverticulitis

SECONDARY OUTCOMES:
conversion to any form of laparoscopy | intraoperative
  conversion to any form of laparoscopy different from peritoneal lavage (with or without bowel resection)
conversion to laparotomy | intraoperative
  conversion to laparotomy (with or without bowel resection)
30 days post-operative mortality | 30 days
30 days post-operative surgical re-interventions rate | 30 days
30 days post-operative percutaneous drainage rate | 30 days
hospital readmission rate for recurrence of diverticulitis | 30 days
visualisation of colonic perforation | intraoperative
  rate of visualisation of colonic perforation during laparoscopic peritoneal lavage
visceral adhesiolysis | intraoperative
  consistency, if any, of visceral adhesiolysis performed during the procedure
duration of follow-up | 12
post-lavage elective resection rate (lavage "bridge" to resection) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gian Andrea Binda, MD, Principal Investigator — Ospedali Galliera, Genova, Italy; Roberto Cirocchi, MD, Principal Investigator — University of Perugia - Terni; Salomone Di Saverio, MD, Principal Investigator — Maggiore Hospital, AUSL Bologna, Italy; Nereo Vettoretto, MD, Principal Investigator — Ospedale Montichiari, Italy
Locations (1):
- Gian Andrea Binda, Genova, Italy

IPD SHARING:
Plan to Share IPD: Yes